CLINICAL TRIAL: NCT02040233
Title: A Double Blinded, Placebo Controlled, Study to Investigate the Safety, Tolerability, Pharmacokinetics and Acute Cardiovascular Responses of a 7 Day Oral Treatment With the Partial Adenosine A1 Receptor Agonist BAY1067197 in Patients With Chronic Systolic Heart Failure: the PARSiFAL-pilot Study.
Brief Title: Multiple Dose Study in Heart Failure of BAY 1067197
Acronym: PARSiFAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16782; 2013-002522-23 (EudraCT Number)
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BAY1067197 (10 mg) (Active Comparator)
  Interventions: Drug: BAY1067197 (10 mg)
- BAY1067197 (Active Comparator)
  Interventions: Drug: BAY1067197
- Placebo (10 mg) (Placebo Comparator)
  Interventions: Drug: Placebo (10 mg)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1067197 (10 mg) — 10 mg BAY1067197 for 7 d treatment once daily as oral application
  Arms: BAY1067197 (10 mg)
Drug: BAY1067197 — The dose escalation to the second dose step will proceed only if the previous dose step has shown acceptable safety and tolerability 5 mg / or 10 mg / or 20 mg BAY1067197 for 7 d treatment as oral application.
  Arms: BAY1067197
Drug: Placebo (10 mg) — 10 mg Placebo for 7 d treatment once daily as oral application
  Arms: Placebo (10 mg)
Drug: Placebo — 5 mg / or 10 mg / or 20 mg Placebo for 7 d treatment once daily as oral application
  Arms: Placebo

SUMMARY:
This is a study to investigate the safety, tolerability and early effects on cardiac function of the partial A1 agonist BAY1067197 in patients with chronic heart failure. BAY1067197 will be applied once daily over 7 days in addition to standard therapy including a beta-blocker. The aim of the study is to assess if a 7 day treatment with BAY1067197 is well tolerated when given on top of standard therapy for heart failure. Furthermore, the study aims to assess if cardiac function improves in the early course of therapy.

ELIGIBILITY:
* Inclusion Criteria:
* Clinical diagnosis of chronic systolic heart failure of ischemic or non-ischemic etiology:(New York Heart Association)NYHA class I-III and treatment with standard pharmacological therapy for the treatment of systolic heart failure including β-blocker ≥ 4 weeks prior to randomization
* Left ventricular ejection fraction ≤ 40%: by any imaging technique within the last 3 months will be accepted for screening purposes but will be verified by baseline CMR(Cardiac Magnetic Resonance Tomography)
* Sinus rhythm for at least 4 weeks prior to randomization
* No planned changes to heart failure related drug therapy for the duration of study drug treatment
* Substantial dysfunctional but viable myocardium as demonstrated by the baseline CMR: Based on a standard 17-segment model (AHA - American Heart Association), 3 or more segments require demonstration of dysfunction (defined by visible assessment of the performing investigator) and viability (defined as < 25% of segment area with scar burden - in patients with CAD (Coronary Artery Disease) or no (i.e. zero) scar burden in patients without CAD [idiopathic CM patient])
* Men or confirmed postmenopausal women or women without childbearing potential.
* Age: 18 to 75 years (inclusive) at the first screening visit.
* Body Mass Index (BMI) :above /equal 18.0 and below/equal 34.9kg/m²
* Exclusion Criteria:
* Atrial fibrillation / atrial flutter within the last 4 weeks prior to randomization or currently persistent/permanent atrial fibrillation / atrial flutter
* Primary valvular disease (severe valvular disease) with planned valve repair or replacement
* Non-idiopathic non-ischemic causes for cardiomyopathy (constrictive, restrictive, or hypertrophic cardiomyopathy; acute myocarditis)
* Listing for heart transplantation and/or anticipated/implanted ventricular assist device Clinically relevant ventricular arrhythmias within the last 2 months (sustained ventricular tachycardia, ventricular flutter or fibrillation), based on either medical history or ICD-testing results (if applicable)
* Unstable cardiac condition, indicated by requirement of IV drug (diuretic, inotrope, etc.) or NYHA IV within 4 weeks prior to randomization
* Coronary revascularization within 4 weeks prior to randomization or if revascularization is anticipated or needed
* Current permanent or intermittent AV-Block > I° or history of AV-Block > I° within six months before enrollment
* PR duration ≥ 300 ms
* Acute Coronary Syndrome (defined as unstable angina [UA], non-ST elevation myocardial infarction [NSTEMI], ST elevation myocardial infarction [STEMI]) within 2 months prior to randomization
* Subjects with untreated hyperthyroidism or hypothyroidism and non-stable thyroid function (intake of stable thyroid hormone substitution allowed)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2015-01-29 (Actual); Study Completion 2015-04-02 (Actual)

PRIMARY OUTCOMES:
Number of Subjects With Relevant Changes in Heart Rate | From the start of study treatment up to Day 29
  Heart rate was measured by monitor measurements after 30 minutes resting in a supine position. The relevant changes in heart rate were recorded and analysed.
Number of Subjects With Relevant Changes in Blood Pressure | From the start of study treatment up to Day 29
  Blood pressure was measured by monitor measurements after 30 minutes resting in a supine position. The relevant changes in blood pressure were recorded and analysed.
Number of Subjects With More than First Degree Atrio-Ventricular (AV) Block | After 7 day tratment and day 28
  A complete standard 12-lead ECG was recorded and evaluated parameters such as heart rate, PR/PQinterval, QRSD interval, QT interval (uncorrected). Clinically relevant findings in ECG such as a second degree AV-block Mobitz type I (Wenkebach), Mobitz type II - or any third-degree AV block were recorded and reported. A 24-hour Holter ECG was recorded with a standard Holter ECG recorder for the purpose of detecting AV blocks, no higher degree AV blocks > 1 or clinically relevant effect on HR were observed during Holter monitoring periods.
Change From Baseline in Left Ventricular Ejection Fraction (LVEF) | Baseline to day 7
  The change in LVEF between the post and the pre-treatment measurements were analyzed using Bayesian statistics to quantify the difference between BAY1067197 treatment and placebo measured by CMR. LVEF is the fraction of blood (in percent) pumped out of the heart's left ventricular chamber with each heart beat, and is a measure of cardiac output for the heart.
Maximum Observed Concentration of BAY84-3174 in Plasma (Cmax) After First Dose of BAY1067197 | Day 1: pre-dose and 0.5, 1, 2, 3, 4, 6, 12 and 24 hours post-dose
  Maximum observed BAY84-3174 concentration in plasma, directly taken from analytical data. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Concentration of BAY84-3174 in Plasma Divided by Dose (Cmax/D) After First Dose of BAY1067197 | Day 1: pre-dose and 0.5, 1, 2, 3, 4, 6, 12 and 24 hours post-dose
  Maximum observed drug concentration, directly taken from analytical data, divided by dose. Geometric mean and %CV were reported.
Area Under the Concentration Versus Time Curve of BAY84-3174 for the Dosing Interval (AUCtau) After First Dose of BAY1067197 | Day 1: pre-dose and 0.5, 1, 2, 3, 4, 6, 12 and 24 hours post-dose
  AUCtau is defined as area under the plasma concentration time profile from time zero to the end of the dosing interval after the first dose and dosing interval was 24 h for both arms. Geometric mean and %CV were reported.
Area Under the Concentration Versus Time Curve of BAY84-3174 for the Dosing Interval Divided by Dose (AUCtau/D) After First Dose of BAY1067197 | Day 1: pre-dose and 0.5, 1, 2, 3, 4, 6, 12 and 24 hours post-dose
  AUCtau/D is defined as area under the plasma concentration time profile from time zero to the end of the dosing interval divided by dose after the first dose and dosing interval was 24 h for both arms. Geometric mean and %CV were reported.
Maximum Observed Concentration of BAY84-3174 in Plasma (Cmax,md) After Multiple Dose Administration During a Dosing Interval | Day 7: pre dose and 0.5, 1, 2, 3, 4, 6 and 12 hours post dose; Day 8, Day 14, Day 22 and Day 29
  Cmax,md is defined as maximum observed drug concentration in plasma after multiple-dose administrations during a dosing interval directly taken from analytical data.Geometric mean and %CV were reported.
Maximum Observed Concentration of BAY84-3174 in Plasma Divided by Dose (Cmax,md/D) After Multiple Dose Administration During a Dosing Interval | Day 7: pre dose and 0.5, 1, 2, 3, 4, 6 and 12 hours post dose; Day 8, Day 14, Day 22 and Day 29
  Maximum observed drug concentration, directly taken from analytical data divided by dose after multiple doses. Geometric mean and %CV were reported.
Area Under the Concentration Versus Time Curve of BAY84-3174 During any Dosing Interval (AUCtau,md) After Multiple Dose Administration | Day 7: pre-dose and 0.5, 1, 2, 3, 4, 6, 12 and 24 hours post-dose
  AUCtau,md is defined as area under the plasma concentration time profile from time zero during the dosing interval after multiple-dose administrations and dosing interval was 24 h for both arms.
  Geometric mean and %CV were reported.
Area Under the Concentration Versus Time Curve of BAY84-3174 During any Dosing Interval Divided by Dose (AUCtau,md/D) After Multiple Dose Administration | Day 7: pre-dose and 0.5, 1, 2, 3, 4, 6, 12 and 24 hours post-dose
  AUCtau,md/D is defined as area under the plasma concentration time profile from time zero to the end of the dosing interval after multiple dose of administrations divided by dose and dosing interval was 24 h for both arms. Geometric mean and %CV were reported.

SECONDARY OUTCOMES:
Changes From Baseline for Wall Motion Score Index at Day (WMSI) as Measured by Cardiac Magnetic Resonance at Day 7 | Baseline to day 7
  Wall motion score index will cover the changes in wall motion score from baseline also.
Number of Subjects With Clinically Relevant Changes Observed in Echocardiography Parameters | Baseline, Day 6 and 15
  Septal mitral annulus (e' septal), Lateral mitral annulus (e' lateral), E/e' average (average of e' lateral and e' septal), E/e' Lateral ratio, E/e' Septal ratio, Peak early doppler transmitral flow velocity (E), Peak atrial doppler transmitral flow velocity (A), E/A Ratio, Deceleration time (DT), Global longitudinal strain, Cardiac output, Stroke volume, Stroke volume index, Peak systolic tissue Doppler Velocity (Smax), Left ventricular end-systolic volume (LVESV), Left ventricular enddiastolic volume (LVEDV), Left atrial volume index (LAVI), Peak pulmonary systolic pressure (PAPsys).
Number of Subjects With Clinically Relevant Changes Observed in Biomarkers | Baseline up to Day 15
  N-terminal prohormone of brain natriuretic peptide (NT-proBNP), renin, mid-region pro-atrial natriuretic peptide (MR-proANP) are biomarkers which show effect on neurohormones.
Time to Reach Maximum Observed Concentration of BAY84-3174 in Plasma (tmax) After First Dose of BAY1067197 | Day 1: pre-dose and 0.5, 1, 2, 3, 4, 6, 12 and 24 hours post-dose
  Time to reach maximum drug concentration in the measured matrix, directly taken from analytical data
Area Under the Concentration Versus Time Curve of BAY84-3174 for the Dosing Interval Divided by Dose per Body Weight (AUCtau,md,norm) After Multiple Dose Administration | Day 7: pre-dose and 0.5, 1, 2, 3, 4, 6, 12 and 24 hours post-dose
  AUCtau,md,norm is defined as area under the plasma concentration time profile from time zero to the end of the dosing interval after multiple dosing divided by dose per body weight. The dosing interval was 24 h for both arms. Geometric mean and %CV were reported.
Maximum Observed Concentration of BAY84-3174 in Plasma Divided by Dose per Body Weight (Cmax,md,norm) After Multiple Dose Administration | Day 7: pre dose and 0.5, 1, 2, 3, 4, 6 and 12 hours post dose; Day 8, Day 14, Day 22 and Day 29
  Cmax,md,norm defined as maximum observed drug concentration in plasma after the first dose followed by multiple-dose administrations during a dosing interval divided by dose per body weight. Geometric mean and %CV were reported.
Time to Reach Maximum Observed Concentration of BAY84-3174 in Plasma (tmax,md) After Multiple Dose Administration | Day 7: pre dose and 0.5, 1, 2, 3, 4, 6 and 12 hours post dose; Day 8, Day 14, Day 22 and Day 29
  tmax,md defines as time to reach maximum drug concentration in the measured matrix after multiple dose administrations directly taken from analytical data.
Half-Life Associated With the Terminal Slope (t1/2,md) After Multiple-Dose Administration | Day 7: pre dose and 0.5, 1, 2, 3, 4, 6 and 12 hours post dose; Day 8, Day 14, Day 22 and Day 29
  t1/2,md is defiend as time to reach maximum observed drug concentration in plasma after the first dose followed by multiple-dose administrations. Geometric mean and %CV were reported.
Maximum Observed Concentration of BAY84-3174 in Plasma After First Dose Divided by Dose per Body Weight (Cmax,norm) | Day 1: pre-dose and 0.5, 1, 2, 3, 4, 6, 12 and 24 hours post-dose
  Cmax,norm is defined as maximum observed drug concentration in plasma after the first dose divided by dose per body weight. Geometric mean and %CV were reported.
Area Under the Concentration Versus Time Curve of BAY84-3174 for the Dosing Interval Divided by Dose per Body Weight (AUCtau,norm) After First Dose of BAY1067197 | Day 1: pre-dose and 0.5, 1, 2, 3, 4, 6, 12 and 24 hours post-dose
  AUCtau,norm is defined as area under the plasma concentration time profile from time zero to the end of the dosing interval divided by dose per body weight after the first dose. Dosing interval was 24 h for both arms. Geometric mean and %CV were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Berlin, Germany
- Italy (3):
  - Bergamo, Lombardy
  - Brescia, Lombardy
  - Milan, Lombardy
- Groningen, Netherlands
- Wroclaw, Poland

REFERENCES:
- See also: Click here and search for information provided by the EMA — http://www.clinicaltrialsregister.eu